CLINICAL TRIAL: NCT04174079
Title: A Prospective, Randomized Controlled Clinical Trial of Adjuvant Chemotherapy After Total Two-field Lymph Node Dissection of Thoracic Esophageal Squamous Cell Carcinoma
Brief Title: Study on Adjuvant Chemotherapy After Total Two-field Lymph Node Dissection of Thoracic Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Peng Lin, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2019-061-01
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Thoracic Esophageal Squamous Cell Carcinoma
Keywords: adjuvant chemotherapy
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): patients with R0 resected T≥3 or N≥1 thoracic esophageal squamous cell carcinoma began to receive chemotherapy of docetaxel combined with nedaplatin within 8 weeks after total two-field lymph node dissection. Docetaxel 75mg/m2 day 1, nedaplatin 75mg/m2 day 1, every 21 days for 4 cycles
  Interventions: Drug: chemotherapy
- control group (No Intervention): patients with R0 resected T≥3 or N≥1 thoracic esophageal squamous cell carcinoma were reviewed regularly after surgery.

INTERVENTIONS:
Drug: chemotherapy — patients with R0 resected T≥3 or N≥1 thoracic esophageal squamous cell carcinoma began to receive chemotherapy of docetaxel combined with nedaplatin within 8 weeks after total two-field lymph node dissection. Docetaxel 75mg/m2 day 1, nedaplatin 75mg/m2 day 1, every 21 days for 4 cycles
  Arms: Experimental group

SUMMARY:
Patients with thoracic esophageal squamous cell carcinoma after total two-field lymph node dissection were randomized into the adjuvant chemotherapy group or the postoperative observation group

DETAILED DESCRIPTION:
Patients with T≥3 or N≥1 thoracic esophageal squamous cell carcinoma after total two-field lymph node dissection were randomly enrolled into the experimental group for adjuvant chemotherapy or the controlled group for postoperative observation. The experimental group received 4-course chemotherapy of docetaxel combined with nedaplatin, and to observe the 3-year progression free survival (DFS) and 5-year overall survival (OS) in two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with esophageal squamous cell carcinoma who received radical surgical resection and total two-field lymph node dissection did not receive neoadjuvant therapy before surgery, and didn't suffer serious complications after surgery.
2. T≥3 or N≥1, and more than 15 lymph nodes were dissected.
3. Age ≥18 years and ≤75 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
5. Adequate hematological function:

   absolute neutrophil count (ANC) ≥ 1.5×109/L, and blood platelet count (PLT) ≥ 1.5×109/L, and hemoglobin ≥ 9g/dL.
6. Adequate hepatic function: total bilirubin ≤1.5 times the upper limit of normal (ULN), aspartate aminotransferase, alanine aminotransferase, and alkaline phosphatase ≤2.5 × ULN.
7. Adequate renal function:

   serum creatinine ≤1.5 × ULN and creatinine clearance ≥50 ml/min.
8. Subjects could understand and comply with study and follow-up procedures, and voluntarily signed written informed consent

Exclusion Criteria:

1. Suffering from previous primary malignancy or co-existing serious illness of other organs, which will affect the judgment of the end point of this study.
2. Serious postoperative complications that will affect progress of chemotherapy.
3. Patients with chemotherapy contraindications.
4. Women who are pregnant or breast-feeding or who are planning for pregnancy.
5. Unable to complete the follow-up as planned.
6. Without informed consent due to psychological, family, social and other factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | At most 5 years after enrollment
  Patients were images with computed tomography (CT) scan

SECONDARY OUTCOMES:
overall survival | At most 5 years after enrollment
  Patients were images with computed tomography (CT) scan

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Uniersity Cancer Center, Guangzhou, Guangdong, China